CLINICAL TRIAL: NCT01731717
Title: Effektivität Und Effizienz Von Behandlungspfaden für Patienten Mit Depressiven Erkrankungen: Stepped Care Als Ansatz für Ein Leitliniengerechtes Und Integriertes Versorgungsmanagement
Brief Title: Cluster Randomized Trial of Stepped Care Intervention vs. Treatment as Usual for Patients With Depression
Acronym: SCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, PD Dr. phil. Birgit Watzke, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01KQ1002B-TP7
Record Dates: First submitted 2012-11-12; First posted 2012-11-22 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Depression
Keywords: depression; stepped care; evidence-based medicine; health services research; psychotherapy; complex intervention; guideline
MeSH Terms: conditions — Depression | interventions — Bibliotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stepped care intervention (SCM) (Experimental): Patients within the stepped care intervention are screened by general physician using the PHQ-9 (inclusion criterion: >4 points) and diagnosed according to International Classification of Diseases (ICD-10) criteria. Patients receive differentially intensive treatment according to depression severity.
  Patients with mild depression receive:
  Step I: Active monitoring or Step II: II.a. Bibliotherapy or II.b. Online self-help ("Deprexis®") or II+: Telephone-based psychotherapy
  Patients with moderate depression receive:
  Step III: III.a. Outpatient psychotherapy or III.b. Psychopharmacological treatment
  Patients with severe depression receive:
  Step IV: Combined psychotherapy and psychopharmacological treatment, optionally in inpatient setting.
  Interventions: Behavioral: Active monitoring; Behavioral: Bibliotherapy; Behavioral: Online self-help; Behavioral: Outpatient psychotherapy; Procedure: Psychiatric treatment; Behavioral: Combined psychotherapy and psychopharmacological treatment
- Control group: treatment as usual (Active Comparator): Patients in the control group are screened by their general physician using the PHQ-D-9 depression scale. Patients included in the study then receive treatment as usual from general physician or other health service providers.
  Interventions: Other: Control group: treatment as usual

INTERVENTIONS:
Behavioral: Active monitoring — General physician performs monitoring every 2 weeks using the PHQ-9 depression scale.
  Arms: Stepped care intervention (SCM)
Behavioral: Bibliotherapy — Patient works with self-help book "Selbsthilfe bei Depressionen" (Görlitz, 2010) under general physician's supervision.
  Arms: Stepped care intervention (SCM)
Behavioral: Online self-help — Patient works with online self-help program "Deprexis" under general physician's supervision.
  Arms: Stepped care intervention (SCM)
Behavioral: Outpatient psychotherapy — Patient receives outpatient psychodynamic or cognitive-behavioural psychotherapy from a psychotherapist participating in the network.
  Arms: Stepped care intervention (SCM)
Procedure: Psychiatric treatment — Patient receives treatment from psychiatrist or general physician participating in the network, this includes psychopharmacotherapy. Treatment takes place within routine care, thus psychiatrists or general physicians individually determine the type of medication and are committed to follow the recommendations of the German S3-Guideline/National Disease Management Guideline for Unipolar Depression.
  Arms: Stepped care intervention (SCM)
Behavioral: Combined psychotherapy and psychopharmacological treatment — Patient receives psychotherapy combined with psychopharmacological treatment, if necessary in inpatient setting.
  Arms: Stepped care intervention (SCM)
Other: Control group: treatment as usual — treatment as usual
  Arms: Control group: treatment as usual

SUMMARY:
The main aim of the project is the implementation and evaluation of a stepped care model (SCM) for patients with depression with 6 treatment options of varying intensity and setting, including innovative technologies (e-mental health, telephone-based psychotherapy). Within this complex intervention, patients are treated by a multiprofessional network of health care providers in Hamburg, Germany. The study compares the SCM condition (intervention group) to a control group receiving treatment as usual (cluster randomization on the level of participating general practitioners). It is expected that the SCM condition will show better results regarding reduction of mental symptoms, improvement of quality of life, more efficient access to care and better cost-benefit ratio.

ELIGIBILITY:
Inclusion Criteria:

* >4 points on PHQ-D-9 depression scale
* sufficient knowledge of German language
* health situation that allows questionnaire completion

Exclusion Criteria:

* insufficient knowledge of German language
* health situation not allowing questionnaire completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in depression severity (PHQ-D-9) | Baseline, 3 months, 6 months, 12 months
  Change in patient-rated depression symptom severity: Patient Health Questionnaire 9, German version (PHQ-D-9; Löwe, Zipfel & Herzog, 2002)

SECONDARY OUTCOMES:
Cost-benefit ratio (QALYs) | Baseline, 6 months, 12 months
  Cost-benefit ratio in quality-adjusted life years(QALYs)
Response/Remission/Relapse (PHQ-D-9) | Baseline, 3 months, 6 months, 12 months
  Response/Remission/Relapse as computed by the difference in pre-post depression severity (PHQ-D-9)
Quality of life (EQ-5D) | Baseline, 3 months, 6 months, 12 months
  Quality of life as measured by EuroQol's EQ-5D
Quality of life (SF-12) | Baseline, 3 months, 6 months, 9 months
  Quality of life as measured by the 12-item Short Form Health Survey (SF-12)
Health service utilization and medication consumption | Baseline, 6 months, 12 months
  Non-standardized items regarding the amount and cost of health services utilized in the past 6 months
Self-esteem | Baseline, 3 months, 6 months, 12 months
  Rosenberg self-esteem scale
Therapeutic alliance | Baseline, 3 months, 6 months, 12 months
  Patient-rated therapeutic alliance as measured by the Helping Alliace Questionnaire (HAQ)
Anxiety symptoms (PHQ-D) | Baseline, 3 months, 6 months, 12 months
  Anxiety as rated by the PHQ-D anxiety scale
Panic symptoms (PHQ-D) | Baseline, 3 months, 6 months, 12 months
  Panic symptoms as measured by the PHQ-D
Somatisation (PHQ-D) | Baseline, 3 months, 6 months, 12 months
  Somatisation as measured by the PHQ-D
General anxiety disorder (GAD-7) | Baseline, 3 months, 6 months, 12 months
  Symptoms of general anxiety disorder measured by the GAD-7

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Watzke, Prof. Dr., Study Director — Centre for Psychosocial Medicine, Department of Medical Psychology, University Medical Centre Hamburg-Eppendorf, Hamburg, Germany; Martin Härter, Prof. Dr. Dr., Study Director — Centre for Psychosocial Medicine, Department of Medical Psychology, University Medical Centre Hamburg-Eppendorf, Hamburg, Germany
Locations (1):
- Centre for Psychosocial Medicine, Department of Medical Psychology, University Medical Centre Hamburg-Eppendorf, Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Brettschneider C, Heddaeus D, Steinmann M, Harter M, Watzke B, Konig HH. Cost-effectiveness of guideline-based stepped and collaborative care versus treatment as usual for patients with depression - a cluster-randomized trial. BMC Psychiatry. 2020 Aug 28;20(1):427. doi: 10.1186/s12888-020-02829-0. PMID 32859177
- [Derived] Watzke B, Heddaeus D, Steinmann M, Konig HH, Wegscheider K, Schulz H, Harter M. Effectiveness and cost-effectiveness of a guideline-based stepped care model for patients with depression: study protocol of a cluster-randomized controlled trial in routine care. BMC Psychiatry. 2014 Aug 20;14:230. doi: 10.1186/s12888-014-0230-y. PMID 25182269